CLINICAL TRIAL: NCT06243458
Title: A Phase II, Open-label, Multicenter Study of Orally Administered RVU120 for the Treatment of Anemia in Patients With Lower-risk Myelodysplastic Neoplasms (MDS)
Brief Title: RVU120 for Treatment of Anemia in Patients With Lower-risk Myelodysplastic Neoplasms
Acronym: (MDS)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GCP-Service International West GmbH (Industry)
Collaborators: Universitätsklinikum Leipzig (Other); Saint-Louis Hospital, Paris, France (Other); University of Florence (Other); University of Salamanca (Other); Medical University of Warsaw (Other); Ryvu Therapeutics SA (Industry); European Myelodysplastic Neoplasms Cooperative Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REMARK_001; EUCT Number 2023-509947-29 (Other: CTIS / EMA)
Record Dates: First submitted 2024-01-25; First posted 2024-02-06 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Low Risk Myelodysplastic Syndromes
Keywords: CDK8/19 Inhibitor; RVU120 (SEL120); Clinical Trial, Phase II

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm RVU120 (Experimental)
  Interventions: Drug: RVU120 (SEL120)

INTERVENTIONS:
Drug: RVU120 (SEL120) — RVU120 will be taken orally every other day (q.o.d). in a 21-day treatment cycle. Doses of RVU120 will be administered from day 1 to day 13 (total of 7 doses per cycle).

SUMMARY:
This study will evaluate orally administered RVU120, a novel small molecule Cyclin-dependent Kinase (CDK) 8/19 inhibitor, in terms of erythroid hematologic improvement (HI-E) and safety in participants with lower-risk myelodysplastic syndrome (MDS). Responding patients are eligible to continue treatment until loss of response/disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided prior to any study-related procedure
2. Age ≥18 years
3. Diagnosis of de novo myelodysplastic neoplasms (MDS) according to World Health Organization (WHO) 2022 criteria.

   Diagnosis will be confirmed during screening assessment.
4. Very low, low or intermediate risk disease MDS with up to 3.5 points according to International Prognostic Scoring System Score Revised (IPSS-R) classification (to be confirmed during screening assessment).

   Patients with del(5q) and max. one further abnormality (excluding monosomy 7, del(7q), TP53mut) are eligible.
5. Symptomatic anemia: Symptomatic anemia (all non transfusion dependent (NTD), low transfusion burden (LTB), or high transfusion burden (HTB)) has to be documented in the 16 weeks baseline period ending on the day of inclusion.

   Patients should be registered only if it is expected at time of registration that
   * a valid and complete Hb (at least five measurements in the period of 16 weeks before the first dose of IMP) and transfusion history will be available at inclusion AND
   * the Hb Mean over the baseline period will be less than 10 g/dL OR three or more red blood cell (RBC)-transfusions will have been given during the baseline period documenting transfusion dependence.
6. No available option of an approved MDS therapy according to decision of the treating physician and based on the following:

   Patients must be
   * ESA exposed (and refractory or intolerant) or ESA naïve and serum erythropoietin level >200 U/L AND/OR
   * Luspatercept exposed (and refractory or intolerant) or luspatercept naïve and not eligible for treatment (e.g. not approved) AND/OR
   * Lenalidomide exposed (and refractory or intolerant) or lenalidomide naïve and not eligible for treatment (e.g. due to non-presence of del(5q))
7. Eastern Cooperative Oncology Group (ECOG) performance score of 0-2
8. Patients must have been off anti-cancer treatment for 2 weeks or 5 half-lives, whichever is longer
9. Clinical laboratory parameters as follows:

   * Peripheral white blood cell (WBC) count, no upper or lower limit at screening, but must be <10 x 109/L prior to first dose of study drug
   * Platelets count >25,000/μL
   * Serum albumin ≥ 30 g/L (3.0 g/dL)
   * Normal coagulation (elevated International Normalized Ratio (INR), prothrombin time or activated partial thromboplastin time (APTT) <1.3 x ULN acceptable)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 x the upper limit of normal (ULN)
   * Total bilirubin ≤1.5 x ULN
   * Creatinine clearance ≥60 mL/min
   * Urine protein < 2+ (as measured by dipstick) or ≤1000 mg/24 hours urine
10. Adequate cardiac function confirmed by left ventricular ejection fraction (LVEF) ≥40% as per echocardiography or MUGA (Multiple Gated Acquisition) scan
11. For females of childbearing potential (FCBP), a negative serum pregnancy test must be confirmed before enrolment. FCBP must commit to use of highly effective method of contraception during study participation and until 28 weeks (6.5 months) after the last dose of study drug. Females must also refrain from donating blood or egg (ovum) during the same time-period.
12. For males, an effective barrier method of contraception must be used during study participation until 28 weeks (6.5 months) after the last dose of study drug, if the patient is sexually active with a FCBP. Males must also refrain from donating blood or sperm during the same time-period.
13. Investigator considers the patient to be suitable for participation in the clinical study by assessing that they:

    * Understand the requirements of the clinical study and can give informed consent.
    * Can comply with study medication dosing requirements and all study-related procedures and evaluations; and
    * Are not considered to be potentially unreliable and/or not cooperative
14. Has received all Coronavirus disease-19 (COVID-19) vaccinations per relevant national guidelines.

Exclusion Criteria:

1. Inability to swallow and retain oral medications.
2. Patient does not accept bone marrow sampling during screening and after the treatment.
3. Prior treatment with azacitidine (injectable or oral) or decitabine.
4. The patient medically requires treatment with the following drugs that are forbidden during the trial or was exposed to one of these 14 days before the first dose of the IMP:

   * Erythropoiesis stimulating agent (ESA) or luspatercept
   * Granulocyte colony-stimulating factor (G-CSF) and granulocyte-macrophage colony stimulating factor (GM-CSF)
   * Lenalidomide
   * Another investigational drug or device, or approved therapy for investigational use
5. Iron chelation therapy NOTE: if therapy was initiated 56 days or more prior to the first dose of the IMP, patient can be included. Recently initiated iron chelation [< 56 days prior to registration] might influence interpretation of hematological response after start of trial medication.
6. Previous treatment with CDK8-targeted therapy(s).
7. Active central nervous system (CNS) involvement.
8. Patients who have undergone major surgery within 28 days prior to first dose of study drug.
9. Evidence of ongoing and uncontrolled systemic bacterial, fungal, or viral infection and acute inflammatory conditions (including pancreatitis)
10. Hematopoietic stem cell transplant within 120 days prior to first dose of study drug.
11. Active Grade 2-4 acute graft versus host disease (GVHD), active moderate-to-severe chronic GVHD, or requirement for systemic immunosuppressive medications for GVHD.
12. Known seropositivity or history of active viral infection with human immunodeficiency virus (HIV).
13. Ongoing significant liver disease such as cirrhosis, drug-induced liver injury, active hepatitis or chronic persistent hepatitis B and/or C:

    * Positive serologic or polymerase chain reaction (PCR) test results for acute or chronic Hepatitis B virus (HBV) infection. Patients whose HBV infection status cannot be determined by serologic test results must be negative for HBV by PCR to be eligible for study participation.
    * Acute or chronic Hepatitis C virus (HCV) infection. Patients who are positive for HCV antibody must be negative for HCV by PCR to be eligible for study participation
14. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RVU120 (e.g. active inflammatory bowel disease, ulcerative disease, malabsorption syndrome, short bowel syndrome, uncontrolled nausea, vomiting or diarrhea).
15. Ongoing drug-induced pneumonitis.
16. Concurrent participation in another investigational clinical trial.
17. Taking any medications, herbal supplements or other substances (including smoking) that are known to be strong inhibitors or moderate/strong inducers or sensitive substrates of CYP1A2, within less than 5 half-lives, prior to first dose of study drug. Any exception should be discussed with the Coordinating Investigator. For clarity, vaping (use of e-cigarettes) is not considered smoking.
18. Significant cardiac dysfunction defined as myocardial infarction within 12 months of first dose of study drug, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled dysrhythmias, or poorly controlled angina.
19. Currently taking drugs that are documented, in the drug package insert, to have a risk of causing prolonged QTc or torsades de pointes (TdP) within 5 half-lives, prior to first dose of study drug.

    Any exception should be discussed with the Coordinating Investigator.
20. Personal or family history of serious ventricular arrhythmia, or QT interval corrected for heart rate (QTc) ≥470 ms.
21. Any other prior or current medical condition, intercurrent illness, surgical history, physical or electrocardiogram (ECG) findings, laboratory abnormalities, or extenuating circumstance (e.g. alcohol or drug addiction) that, in the Investigator's opinion, could jeopardize patient safety or interfere with the objectives of the study.
22. Prior history of malignancies other than Acute myeloid leukemia (AML) or MDS, unless the patient has been free of the disease for 5 years or more prior to screening. Exceptions to the ≥5-year time limit include history of the following:

    * basal cell carcinoma of the skin
    * non-metastatic squamous cell carcinoma of the skin
    * carcinoma in situ of the cervix
    * carcinoma in situ of the breast
    * carcinoma in situ of the bladder
    * incidental histological finding of prostate cancer (Tumor/Node/Metastasis [TNM] stage of T1a or T1b).
23. Pregnant or breast-feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Erythroid Response (HI-E) Rate of Participants after Treatment with RVU120 (dose of 150 mg) | Response Assessment measured after 8 full Cycles of RVU120 administration. Each cycle is 21 days.
  The International Working Group (IWG) 2018 Hematologic Improvement Criteria for MDS will be used to define responders.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, Prof., Principal Investigator — Universitätsklinikum Leipzig; Lionel Adès, Prof., Principal Investigator — Service d'hématologie seniors Hôpital Saint-Louis, Paris; Valeria Santini, Prof., Principal Investigator — University of Careggi, Italy; Krzysztof Mądry, Dr., Principal Investigator — Medical University of Warsaw; Diez Campelo, Dr., Principal Investigator — University of Salamanca
Locations (25):
- France (5):
  - CHU Grenoble Alpes - Hôpital Michallon, Grenoble
  - CHU de Nice - Hôpital l'Archet 1, Nice
  - Hôpital Saint-Louis, Service d'Hématologie Séniors, Paris
  - CHU de Bordeaux - Centre François Magendie - Groupe Hospitalier Sud, Pessac
  - CHU de Toulouse - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
- Germany (3):
  - Marien Hospital Düsseldorf, Düsseldorf
  - Universität Leipzig, Med. Fak., Klinik und Poliklinik für Hämatologie, Zelltherapie, Hämostaseologie und Infektiologie, Leipzig
  - Universitätsklinikum Münster (UKM), Münster
- Italy (6):
  - AOU delle Marche, Ancona
  - AOU Consorziale Policlinico, Università degli Studi Aldo Moro, Bari
  - Candiolo Cancer Institute, IRCCS Fondazione del Piemonte per l'Oncologia, Candiolo
  - AOU Careggi, Florence
  - IRCCS Humanitas Research Hospital, Milan
  - Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli, Reggio Calabria
- Poland (5):
  - Samodzielny Publiczny Szpital Kliniczny im.Andrzeja Mielęckiego Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Pratia Hematologia Sp. z o. o. , Pratia Onkologia Katowice, Katowice
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M.Kopernika w Łodzi, Lodz
  - MTZ Clinical Research powered by Pratia, Warsaw
  - Uniwersytecki Szpital Kliniczny im.Jana Mikulacza-Radeckiego, Wroclaw
- Spain (6):
  - Hematology Department Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - Hospital Universitario de León, León
  - Hospital Universitario La Paz, Madrid
  - Navarra university clinic, Pamplona
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario de Valencia, Valencia